CLINICAL TRIAL: NCT02761278
Title: Expression of HOXA10 and HOXA11 in the Endometrium of Infertility Patients With an Endometrial Polyp Before and After Polypectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYMC-0039-16
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HOXA10 and HOXA11 Expression Before Polypectomy (Active Comparator): A biopsy will taken in infertility patients with endometrial polyp before polypectomy
  Interventions: Procedure: Endometrial biopsy
- HOXA10 and HOXA11 Expression After Polypectomy (Active Comparator): A biopsy will taken in infertility patients with endometrial polyp 1-3 months after polypectomy
  Interventions: Procedure: Endometrial biopsy

INTERVENTIONS:
Procedure: Endometrial biopsy

SUMMARY:
The aim of this study is to measure the expression of HOXA10 and HOXA11 in the endometrium of infertility patients with an endometrial polyp before and after polypectomy. HOXA10 and HOXA11 are well-established markers of implantation. It is uncertain as to whether an endometrial polyp interferes with embryo implantation. A higher expression of HOXA10 and HOXA11 after polypectomy can indicate that endometrial polyp does interfere with embryo implantation.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women with endometrial polyp

Exclusion Criteria:

* Endometriosis
* Polycystic ovary syndrome
* Hydrosalpinx
* Sub-mucus myoma
* Women who have taken hormonal therapy in the preceding month

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of amounts of HOXA10 and HOXA11 expressed before and after polypectomy | Four months

CONTACTS AND LOCATIONS:
Overall Officials: Guy Shrem, MD, Principal Investigator — Hillel Yaffe Medical Center

IPD SHARING:
Plan to Share IPD: No